CLINICAL TRIAL: NCT04017234
Title: The Effects of Frequency Following Response, Eye Exercise, and Transcutaneous Electrical Nerve Stimulation on Prevention of Myopia Progression in Taiwan Schoolchildren
Brief Title: Eye Exercise, Transcutaneous Electrical Nerve Stimulation on Prevention of Myopia Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CMUH107-REC1-124
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMP group (Experimental): children received health education for eye and the intervention(which included frequency following response, eye exercise, and transcutaneous electrical nerve stimulation) a 30 minute three times per week for four weeks.
  Interventions: Other: frequency following response, eye exercise, and transcutaneous
- control group (No Intervention): children just received health education for eye

INTERVENTIONS:
Other: frequency following response, eye exercise, and transcutaneous — frequency following response, eye exercise, and TENS for 3 times per week during 4 weeks
  Arms: PMP group

SUMMARY:
In Taiwan, the increasing prevalence of myopia shows a decline with age. Myopia has become a serious ocular problem in children because high myopia may lead to retinal damage, cataract and glaucoma. A prevention of myopia progression (PMP) will be developed and examined. This promotion program includes strategies such as a frequency following response, eye exercise, and transcutaneous electrical nerve stimulation on the prevention of myopia progression. Eye exercise defined as a computerized image led motion. The study aims to examine the effect of the implementation on the PMP.

DETAILED DESCRIPTION:
This is an experimental study. A sample size of 25~40 participants from an elementary school will be recruited in the randomized controlled study.The sequential arrangement is arranged in a random manner for the participating children. A investigation of four groups will be designed for the PMP: Group 1 (frequency following response, Group 2(frequency following response,and eye exercise), Group 3 (frequency following response, eye exercise, transcutaneous electrical nerve stimulation and stimulating auricular acupoints), and Group 4, the control group. The PMP implement a 30 minute intervention two times per the investigators. Pre-test and post-test (eyeball diopter detection and Sellen's vision chart) will be carried out. The duration of each intervention is provided for two days. The washout period following next intervention is 7 days at least. After completing four intervention, the effect of the best intervention of eight the investigator will be conducted.The evaluation time of the interventions will be observed at first-time and one-month observations. A descriptive and inferential statistics by SpSS will be used for data analysis.

The investigators will apply the frequency following response, eye exercise, and transcutaneous electrical nerve stimulation on PMP among Taiwan schoolchildren. The findings of the study may provide information for promotion of visual health for schoolchildren and their parents.

ELIGIBILITY:
Inclusion Criteria:

* myopia is defined as the equivalent spherical surface degree of any one is less than or equal to -0.50D
* do not use cyclogel or atropine
* At least the eye ointment is deactivated for at least seven days
* no plastic tablets are currently used
* at least the plastic tablets are not allowed to be retired for more than seven days

Exclusion Criteria:

* Children with current traumatic and unrecoverable other eye disease

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
eyeball structure | one month detection after intervention
  eyeball diopter detection

SECONDARY OUTCOMES:
vision check | one month detection after intervention
  Sellen's vision chart

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kuei Teng, Principal Investigator — China Medical University, Taiwan
Locations (1):
- Chen Pin elementary school, Taichung, Taiwan